CLINICAL TRIAL: NCT07022353
Title: Ultrasound-guided Bi-level Erector Spinae Plane Block and Pre-emptive Single-dose Oral Tizanidine for Postoperative Analgesia After Mastectomy Surgery: a Prospective, Randomized, Controlled Trial
Brief Title: Bi-level Erector Spinae Plane Block and Pre-emptive Oral Tizanidine for Analgesia After Mastectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amany Hazem abdelmaksood EL-deeb, principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP plus oral tizanidine
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Mastectomy Patient
Keywords: Mastectomy; Analgesia; erector spinae plane block; tizanidine
MeSH Terms: conditions — Agnosia | interventions — tizanidine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation, prepare all injections and oral medication needed for the study. Another investigator blinded to the study group will give oral drug and perform block. In addition, the study subjects and the resident assessing the outcome will be blinded to the study group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilevel ESP block group (Active Comparator): patients will have bilevel ESP block plus oral placebo capsule.
  Interventions: Procedure: Bilevel erector spinae plane block; Drug: Placebo Oral Capsule
- Bilevel ESP block + tizanidine group (Active Comparator): patients will have bilevel ESP block plus oral tizanidine capsule.
  Interventions: Procedure: Bilevel erector spinae plane block; Drug: tizanidine oral capsule

INTERVENTIONS:
Procedure: Bilevel erector spinae plane block — Block will be performed unilaterally with the patient in the sitting position leaning forward. The block will be done using a high frequency linear probe (6-13 MHz). The block area will be adequately sterilized and draped, then the ultrasound probe will be placed 2-3 cm laterally from the midline at the level of the T3 spinous process using a sagittal approach to identify the hyperechoic transverse process shadow deep to the trapezius, rhomboid major, and erector spinae muscles. Then, the needle will be inserted craniocaudally in-plane to reach the transverse process deep to the erector spinae muscle. Correct positioning of the needle will be confirmed through real-time visualization of 2-mL saline hydro dissection. After confirmation of needle position, 15 mL of bupivacaine 0.25% will be injected at each level. The same procedure was repeated for the second level T5 spinous process. block failure defined as the presence of full sensation after 30 minutes, patients will be excluded .
  Other Names: ESP
Drug: Placebo Oral Capsule — One hour prior to anesthesia induction, the patients will recieve oral placebo capsule that will have the same color, smell, and size as tizanidine.
  Other Names: Placebo
  Arms: Bilevel ESP block group
Drug: tizanidine oral capsule — One hour prior to anesthesia induction, the tizanidine group will receive a 4 mg tizanidine oral capsule.
  Other Names: tizanidine
  Arms: Bilevel ESP block + tizanidine group

SUMMARY:
Effective management of postoperative pain in breast cancer surgery is essential to minimize the risk of developing postmastectomy pain syndrome.The aim of this study is to evaluate the effectiveness of combining bilevel erector spinae plane (ESP) block with a single preoperative oral dose of tizanidine in improving postoperative analgesia in patients undergoing mastectomy surgery.

It is hypothesized that the combination of bilevel ESP block and single-dose oral tizanidine will provide superior postoperative analgesia compared to bilevel ESP block alone in patients undergoing mastectomy.

DETAILED DESCRIPTION:
Introduction:

Effective management of postoperative pain in breast cancer surgery is essential to minimize the risk of developing postmastectomy pain syndrome, a chronic condition that significantly impacts patients' quality of life. Multimodal analgesia, which combines pharmacological and non-pharmacological strategies, has been shown to enhance postoperative pain control and reduce opioid consumption. In recent years, regional anesthesia techniques have become increasingly favored for perioperative pain management in breast surgeries. The ESP block has gained popularity due to its simplicity, safety profile, and effectiveness in thoracic and breast surgeries. Its analgesic action is attributed to the craniocaudal spread of local anesthetic into the costovertebral foramina and epidural space, resulting in blockade of both ventral and dorsal rami of the spinal nerves and providing unilateral thoracic analgesia.The bilevel ESP block, which involves administering the block at two distinct thoracic levels, has been proposed to enhance the spread of local anesthetic and improve analgesic coverage, particularly in the anterolateral chest wall and axillary regions commonly involved in mastectomy.

Tizanidine has been shown to reduce perioperative opioid and anesthetic requirements, stabilize hemodynamic responses to tracheal intubation, and minimize postoperative complications such as shivering and myocardial ischemia. Previous studies have demonstrated its effectiveness in reducing postoperative pain across a variety of surgical procedures, including laparoscopic cholecystectomy, thyroidectomy, anorectal surgery, hernia repair, and orthognathic surgery.Given the potential synergistic effects of combining regional anesthesia with systemic analgesics, this study aims to evaluate the efficacy of combining bilevel ESPB with a single oral dose of tizanidine for postoperative pain control in patients undergoing mastectomy.

Aim of the Study:

The aim of this study is to evaluate the effectiveness of combining bilevel erector spinae plane (ESP) block with a single preoperative oral dose of tizanidine in improving postoperative analgesia in patients undergoing mastectomy surgery.

Sample Size Calculation:

Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 3.1.9.2 for windows (2017). The primary outcome will be time to first analgesic request. In a pilot study performed on 10 patients using bilevel ESP block, the mean (SD) of time to first analgesic request was 21 (6.5) hours. Using a two-sided hypothesis test with a significance level of 0.05, assuming alpha = 0.05 and beta = 0.2 (power = 80%) and using a two-sided two-sample unequal-variance t-test, 39 subjects will be required in each group to detect 20 % difference between groups which is considered the minimal clinically important difference. To allow for subject dropouts, 45 subjects will be assigned to each group.

Methods; The study will be conducted in Mansoura oncology centre on 90 patients who will be scheduled for mastectomy surgery under general anesthesia. Informed written consent will be obtained from all subjects in the study after ensuring confidentiality. 90 eligible patients will be randomly assigned to 2 equal groups (Bilevel ESP block group) and (Bilevel ESP block+ tizanidine group) according to computer-generated table of random numbers using the permuted block randomization method. The group allocation will be concealed in sequentially numbered, sealed opaque envelopes which will be opened only after obtaining the written informed consent.

The study protocol will be explained to all patients along with VAS after enrollment into the study. They will be kept fasting according to pre-operative ASA recommendations prior to surgery. Basic demographic characters including age, gender, and BMI will be recorded.

The peri-operative management will be identical in both groups. All patients with planned modified radical mastectomy will be assessed preoperatively by detailed medical history taking, clinical examination, Electrocardiography (ECG), and basal laboratory investigations as complete blood count (CBC), coagulation profile (PT, INR), blood glucose level, liver and renal function tests (liver enzymes, serum bilirubin, albumin and serum creatinine).

Statistical Methods:

The collected data will be coded, processed, and analyzed using SPSS program (version 22) for Windows. Normality of numerical data distribution will be tested by Shapiro-Wilk test. Continuous data of normal distribution will be presented as mean ± SD and will be compared with the unpaired student's t test. Non-normally distributed data will be presented as median (range) and will be compared with the Mann-Whitney U test. Categorical data will be presented as number (percentage) and will be compared with the Chi-square test. All data will be considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiology (ASA) ІІ patients.
2. Scheduled for unilateral modified radical mastectomy.
3. BMI levels between 18.5- 35 Kg/m2.

Exclusion Criteria:

1. Patient's refusal.
2. Altered mental status or un-cooperative patients.
3. History of known sensitivity to the used anesthetics.
4. Bleeding or coagulation diathesis.
5. Infection or redness at the injection site.
6. Cardiac, renal, hepatic, hematological disease, peptic ulcer, gastrointestinal bleeding, and central or peripheral neurological disease.
7. Chronic pain.
8. Participants used analgesics routinely within the last 24 h.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 90 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
First analgesic request | Up to 24 hours after the procedure.
  The time of the first analgesic request for fentanyl will be recorded.

SECONDARY OUTCOMES:
Visual analogue score (VAS) for pain assessment | Up to 24 hours after the procedure
  VAS score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain) will be assessed before the procedure, and then at 2, 4, 6, 12, and 24 h post operative.
Total analgesic requirements of fentanyl | Up to 24 hours after the procedure
  The amount of fentanyl consumption given as a rescue analgesia to patients will be measured all over the 24 hours.
Heart rate (HR) | Up to the end of the procedure
  HR will be recorded before the procedure, after 15 min, 30 minutes and then every 30min intraoperative till the end of surgery.
Mean arterial blood pressure (MAP) | Up to the end of the procedure
  MAP will be recorded before the procedure, after 15 min, 30 minutes and then every 30min intraoperative till the end of surgery.
Adverse effects | Up to 24 hours after the procedure]
  respiratory depression, bradycardia, hypotension, nausea, vomiting, hematoma or allergic reactions will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Amany H ELDeeb, MD, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Oncology Centre, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yazicioglu D, Caparlar C, Akkaya T, Mercan U, Kulacoglu H. Tizanidine for the management of acute postoperative pain after inguinal hernia repair: A placebo-controlled double-blind trial. Eur J Anaesthesiol. 2016 Mar;33(3):215-22. doi: 10.1097/EJA.0000000000000371. PMID 26555871
- [Background] Woodworth GE, Ivie RMJ, Nelson SM, Walker CM, Maniker RB. Perioperative Breast Analgesia: A Qualitative Review of Anatomy and Regional Techniques. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):609-631. doi: 10.1097/AAP.0000000000000641. PMID 28820803
- [Background] Mohammadi F, Marashi M, Tavakoli I, Khakbaz O. Effects of oral clonidine premedication on hemodynamic status in bimaxillary orthognathic surgery: A double-blind randomized clinical trial. J Craniomaxillofac Surg. 2016 Apr;44(4):436-9. doi: 10.1016/j.jcms.2016.01.004. Epub 2016 Jan 11. PMID 26874557
- [Background] Maniker RB, Damiano J, Ivie RMJ, Pavelic M, Woodworth GE. Perioperative Breast Analgesia: a Systematic Review of the Evidence for Perioperative Analgesic Medications. Curr Pain Headache Rep. 2022 Apr;26(4):299-321. doi: 10.1007/s11916-022-01031-z. Epub 2022 Feb 23. PMID 35195851
- [Background] Kurdi MS, Agrawal P, Thakkar P, Arora D, Barde SM, Eswaran K. Recent advancements in regional anaesthesia. Indian J Anaesth. 2023 Jan;67(1):63-70. doi: 10.4103/ija.ija_1021_22. Epub 2023 Jan 21. PMID 36970484
- [Background] Guan HY, Yuan Y, Gao K, Luo HX. Efficacy and safety of erector spinae plane block for postoperative analgesia in breast cancer surgery-A systematic review and meta-analysis. J Surg Oncol. 2023 May;127(6):905-920. doi: 10.1002/jso.27221. Epub 2023 Feb 24. PMID 36826370
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Elsabeeny WY, Fahmy RM, Elshamy FH, Shehab NN, Abed SM, Taha WS, Ibrahim MA, Gad AF. Role of bilevel erector spinae with high thoracic block vs conventional unilevel block in analgesia and reduction of pain in axilla in breast cancer surgeries: a randomized controlled trial. Pain Rep. 2025 Jan 13;10(1):e1234. doi: 10.1097/PR9.0000000000001234. eCollection 2025 Feb. PMID 39816904
- [Background] Dadmehr S, Shooshtari Z, Alipour M, Eshghpour M, Shaban B, Vaezi T, Samieirad S. Is Preemptive Oral Tizanidine Effective on Postoperative Pain Intensity after Bimaxillary Orthognathic Surgery? A Triple-Blind Randomized Clinical Trial. World J Plast Surg. 2022 Jul;11(2):37-45. doi: 10.52547/wjps.11.2.37. PMID 36117905
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Gumus Demirbilek S. Bi-level erector spinae plane block for the control of severe back pain related to vertebral metastasis. BMJ Case Rep. 2019 Jun 20;12(6):e228129. doi: 10.1136/bcr-2018-228129. PMID 31227568
- [Background] Aksu C, Kus A, Yorukoglu HU, Tor Kilic C, Gurkan Y. Analgesic effect of the bi-level injection erector spinae plane block after breast surgery: A randomized controlled trial. Agri. 2019 Jul;31(3):132-137. doi: 10.14744/agri.2019.61687. PMID 31736025
- [Background] Ahiskalioglu A, Yayik AM, Oral Ahiskalioglu E, Dostbil A, Doymus O, Karadeniz E, Ari MA, Sengoz F, Alici HA, Celik EC. Ultrasound-guided bilateral superficial cervical block and preemptive single-dose oral tizanidine for post-thyroidectomy pain: a randomized-controlled double-blind study. J Anesth. 2018 Apr;32(2):219-226. doi: 10.1007/s00540-018-2468-x. Epub 2018 Feb 21. PMID 29468508